CLINICAL TRIAL: NCT03271281
Title: PET/CT Imaging of Angiogenesis in Patients With Neuroendocrine Tumors Using 68Ga-NODAGA-E[c(RGDyK)]2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Esben Carlsen, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK2017-2; 2017-002512-14 (EudraCT Number)
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Neuroendocrine Tumors
Keywords: 68Ga-NODAGA-E[c(RGDyK)]2; Angiogenesis PET/CT; Neuroendocrine tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Angiogenesis PET/CT (Experimental): One injection of the radioligand 68Ga-NODAGA-E[c(RGDyK)]2 followed by PET/CT
  Interventions: Drug: One injection of 68Ga-NODAGA-E[c(RGDyK)]2; Device: PET/CT

INTERVENTIONS:
Drug: One injection of 68Ga-NODAGA-E[c(RGDyK)]2 — One injection of 68Ga-NODAGA-E[c(RGDyK)]2
Device: PET/CT — Following injection of 68Ga-NODAGA-E[c(RGDyK)]2 the patients will be subjected to whole body PET/CT

SUMMARY:
The aim of this non-randomised, prospective study is to investigate the applicability and prognostic value of angiogenesis PET/CT with the radioligand 68Ga-NODAGA- E[c(RGDyK)]2 in patients with neuroendocrine tumors (NETs).

DETAILED DESCRIPTION:
The radioligand 68Ga-NODAGA- E[c(RGDyK)]2 targets the Arg-Gly-Asp (RGD) sequence known to bind with the αvβ3 integrin that is expressed on the surface of angiogenic blood vessels or tumor cells. The radioligand can be used to visualize tumor angiogenesis using PET/CT.

A total of 120 NET patients will be subjected to an angiogenesis-PET/CT scan. Follow-up will be performed (from the time of the angiogenesis PET/CT) at 6 months for disease specific survival (DSS) and a 1 year follow-up for PFS and OS. The uptake of 68Ga-NODAGA-E[c(RGDyK)]2 (Standardized Uptake Values, SUVmax) in tumor lesions will be quantified as Standardized Uptake Values (SUVmax/SUVmean) and compared with PFS, DSS and OS (dichotomized above/below median SUVmax and analyzed by Kaplan-Meier).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gastro-entero-pancreatic Neuroendocrine Tumors (GEP-NET; grade: G1-G3) or broncho-pulmonary NET.
* WHO performance status 0-2
* Must be able to read and understand the patient information in Danish and to give informed consent

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Weight more than the maximum weight limit for the PET/CT bed of the scanner (140 kg)
* History of allergic reaction attributable to compounds of similar chemical or biologic composition to 68Ga-NODAGA-E[c(RGDyK)]2
* In case of broncho-pulmonary NET, the subtype must not be small cell lung cancer (SCLC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Angiogenesis PET/CT imaging of patients with neuroendocrine tumors | 1 hour
  The radioligand 68Ga-NODAGA-E[c(RGDyK)]2 can be used to visualize neuroendocrine tumors (grade G1-G3)

SECONDARY OUTCOMES:
Angiogenesis PET/CT progonostic factor for progression free survival | 12 months
  The uptake of the 68Ga-NODAGA-E[c(RGDyK)]2 in neuroendocrine tumor lesions (quantified as Standard Uptake Values) is associated with progression free survival (PFS) neuroendocrine tumors (grade G1-G3)
Angiogenesis PET/CT prognostic factor for overall and disease specific survival | 12 months
  The uptake of the 68Ga-NODAGA-E[c(RGDyK)]2 in neuroendocrine tumor lesions (quantified as Standard Uptake Values) is associated with overall and disease specific free survival (PFS) neuroendocrine tumors (grade G1-G3)
Target validation of angiogenesis PET/CT | 2 weeks
  Uptake of 68Ga-NODAGA-E[c(RGDyK)]2 correlates directly to gene expression of angiogenesis markers αvβ3 integrin and VEGF-A in tumor tissue obtained by biopsies or planned surgery (<2 weeks before/after angiogenesis PET/CT)

CONTACTS AND LOCATIONS:
Overall Officials: Esben Carlsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark